CLINICAL TRIAL: NCT02403531
Title: A Phase II Randomized Trial of Induction Chemotherapy Versus no Induction Chemotherapy Followed by Definitive Chemoradiotherapy in Patients With Inoperable Thoracic Esophageal Cancer
Brief Title: Induction Chemotherapy Followed by Chemoradiotherapy in Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mian XI (Other)
Responsible Party: Sponsor-Investigator, Mian XI, Dr. Xi, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICCRTEC
Record Dates: First submitted 2015-03-19; First posted 2015-03-31 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Neoplasms
Keywords: Esophageal cancer; Chemoradiotherapy; induction chemotherapy
MeSH Terms: conditions — Neoplasms; Esophageal Neoplasms | interventions — Docetaxel; Cisplatin; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiotherapy (Active Comparator): Patients assigned to this Arm received concurrent chemoradiotherapy. The prescribed dose of radiotherapy is generally 50-60 Gy/25-28fr. The concomitant chemotherapy is docetaxel 20 mg/m2 on day 1, cisplatin 25 mg/m2 on day 1, repeated weekly during radiation.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: Radiotherapy
- Induction chemotherapy plus chemoradiotherapy (Experimental): Patients assigned to this Arm first received two cycles of 3-weekly schedule of IC before definitive chemoradiotherapy, consisting of docetaxel 75 mg/m2 on day 1 and cisplatin 75 mg/m2 on day 1. The prescribed dose of radiotherapy is generally 50-60 Gy/25-28fr. The concomitant chemotherapy is docetaxel 20 mg/m2 on day 1, cisplatin 25 mg/m2 on day 1, repeated weekly during radiation.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Docetaxel — Include brand names, serial numbers and code names to improve search results on the ClinicalTrials.gov web site.
  Other Names: taxotere
Drug: Cisplatin — Include brand names, serial numbers and code names to improve search results on the ClinicalTrials.gov web site.
  Other Names: DDP
Radiation: Radiotherapy — definitive radiotherapy
  Other Names: radiation

SUMMARY:
The contribution of induction chemotherapy before definitive chemoradiotherapy is unknown. The purpose of this study was to compare the efficacy and toxicity of induction chemotherapy followed by definitive chemoradiotherapy versus no induction chemotherapy in patients with inoperable thoracic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
108 patients were randomized to receive no induction chemotherapy (IC, Arm A) or IC (Arm B) before definitive chemoradiotherapy in patients with inoperable thoracic esophageal squamous cell carcinoma. Patients assigned to Arm B first received two cycles of 3-weekly schedule of IC, consisting of docetaxel 75 mg/m2 on day 1 and cisplatin 75 mg/m2 on day 1. The prescribed dose of radiotherapy is generally 50-60 Gy/25-28fr. The concomitant chemotherapy is docetaxel 20 mg/m2 on day 1, cisplatin 25 mg/m2 on day 1, repeated weekly during radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Localized, nonmetastatic disease (T1-4, N0-1) confirmed by endoscopic ultrasound (EUS) and CT scan (according to UICC TNM version 6);
3. Absence of distant metastasis of solid organ;
4. Not suitable for surgery (either for medical reasons or patient's choice);
5. Age at diagnosis 18 to 70 years;
6. Eastern Cooperative Oncology Group performance status ≤ 2
7. No prior cancer therapy;
8. No history of concomitant or previous malignancy;
9. Hematologic function: WBC ≥ 4.0×109/L, PLT ≥ 80×109/L, Hb ≥ 10mg/dL;
10. Renal function: Cr ≤ 1.25×UNL;
11. Hepatic function: BIL ≤ 1.5×UNL, ALT/AST ≤ 2.5×UNL;
12. Documented informed consent to participate in the trial.

Exclusion Criteria:

1. Younger than 18 or older than 70 years of age;
2. ECOG performance status of 3 or above;
3. Other cancer history;
4. Previous radiotherapy history;
5. Subjects with distant metastases;
6. Pregnancy or breast feeding. Women of childbearing age must use effective contraception;
7. Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension);
8. Evidence of bleeding diathesis or serious infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
overall response rate (clinical complete response and partial response) | 3 months after chemoradiotherapy (plus or minus 7 days)
  RECIST (Response Evaluation Criteria in Solid Tumors) criteria was used to determine the tumor response. Tumor response was evaluated 3 months after the completion of treatment based on barium esophagography, CT scans, and endoscopy with biopsies.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Three years follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Progression-free survival | 3 years
  From the date of randomization to the date of disease progression or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Zhong Liu, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ruhstaller T, Widmer L, Schuller JC, Roth A, Hess V, Mingrone W, von Moos R, Borner M, Pestalozzi BC, BalmerMajno S, Koberle D, Terraciano L, Schnider A, Bodis S, Popescu R; Swiss Group for Clinical Cancer Research (SAKK). Multicenter phase II trial of preoperative induction chemotherapy followed by chemoradiation with docetaxel and cisplatin for locally advanced esophageal carcinoma (SAKK 75/02). Ann Oncol. 2009 Sep;20(9):1522-1528. doi: 10.1093/annonc/mdp045. Epub 2009 May 22. PMID 19465425
- [Background] Koo DH, Park SI, Kim YH, Kim JH, Jung HY, Lee GH, Choi KD, Song HJ, Song HY, Shin JH, Cho KJ, Yoon DH, Kim SB. Phase II study of use of a single cycle of induction chemotherapy and concurrent chemoradiotherapy containing capecitabine/cisplatin followed by surgery for patients with resectable esophageal squamous cell carcinoma: long-term follow-up data. Cancer Chemother Pharmacol. 2012 Mar;69(3):655-63. doi: 10.1007/s00280-011-1750-5. Epub 2011 Oct 4. PMID 21968953
- [Background] Ilson DH, Minsky BD, Ku GY, Rusch V, Rizk N, Shah M, Kelsen DP, Capanu M, Tang L, Campbell J, Bains M. Phase 2 trial of induction and concurrent chemoradiotherapy with weekly irinotecan and cisplatin followed by surgery for esophageal cancer. Cancer. 2012 Jun 1;118(11):2820-7. doi: 10.1002/cncr.26591. Epub 2011 Oct 11. PMID 21990000
- [Background] Ajani JA, Xiao L, Roth JA, Hofstetter WL, Walsh G, Komaki R, Liao Z, Rice DC, Vaporciyan AA, Maru DM, Lee JH, Bhutani MS, Eid A, Yao JC, Phan AP, Halpin A, Suzuki A, Taketa T, Thall PF, Swisher SG. A phase II randomized trial of induction chemotherapy versus no induction chemotherapy followed by preoperative chemoradiation in patients with esophageal cancer. Ann Oncol. 2013 Nov;24(11):2844-9. doi: 10.1093/annonc/mdt339. Epub 2013 Aug 23. PMID 23975663
- [Derived] Liu S, Chen B, Zhu Y, Wang S, Cheng X, Wang R, Hu Y, Liu H, Li Q, Zhang L, Zhao L, Liu M, Xi M. Induction chemotherapy plus chemoradiotherapy in esophageal cancer: long-term results and exploratory analyses of a randomized controlled trial. Oncologist. 2025 Jul 4;30(7):oyae295. doi: 10.1093/oncolo/oyae295. PMID 39584557
- [Derived] Liu S, Luo L, Zhao L, Zhu Y, Liu H, Li Q, Cai L, Hu Y, Qiu B, Zhang L, Shen J, Yang Y, Liu M, Xi M. Induction chemotherapy followed by definitive chemoradiotherapy versus chemoradiotherapy alone in esophageal squamous cell carcinoma: a randomized phase II trial. Nat Commun. 2021 Jun 29;12(1):4014. doi: 10.1038/s41467-021-24288-1. PMID 34188053